CLINICAL TRIAL: NCT00710424
Title: A Double Blind, Randomized, Placebo Controlled, Parallel Group Study of Sativex in the Treatment of Subjects With Pain Due to Diabetic Neuropathy
Brief Title: A Study of Sativex® for Pain Relief Due to Diabetic Neuropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: GWCL0305
Record Dates: First submitted 2008-07-02; First posted 2008-07-04 (Estimated); Results first posted 2012-07-31 (Estimated); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Pain; Diabetic Neuropathy
Keywords: Pain; diabetic neuropathy
MeSH Terms: conditions — Pain; Diabetic Neuropathies | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sativex (Experimental)
  Interventions: Drug: Sativex
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sativex — containing THC (27 mg/ml):CBD (25 mg/ml), in ethanol:propylene glycol (50:50) excipients, with peppermint oil (0.05%) flavouring. Maximum permitted dose was eight actuations in any three hour period and 24 actuations (THC 65 mg: CBD 60 mg) in 24 hours
  Other Names: GW-1000-02
  Arms: Sativex
Drug: Placebo — containing peppermint oil, 0.05% (v/v), quinoline yellow, 0.005% (w/v), sunset yellow, 0.0025% (w/v), in ethanol:propylene glycol (50:50) excipient.
  Other Names: GW-4001-01
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of Sativex® compared with placebo in relieving pain due to Diabetic Neuropathy.

DETAILED DESCRIPTION:
This was a 15 week (one week baseline and fourteen weeks treatment period), multicentre, double blind, randomised, placebo controlled, parallel group study to evaluate the efficacy of Sativex in subjects with pain due to diabetic neuropathy. Subjects were screened to determine eligibility and completed a seven-day baseline period. Subjects then returned to the centre for assessment, randomisation and dose introduction. Visits occurred at the end of weeks two, six, ten and at the end of the study (treatment week 14) or earlier if they withdrew. A follow up visit occurred 28 days after completion or withdrawal. Subjects in this study were given the opportunity to be enrolled in an open label extension study.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent.
* Male or female, aged 18 years or above.
* Ability (in the investigators opinion) and willingness to comply with all study requirements.
* Diagnosed with Type 1 or 2 diabetes mellitus as diagnosed according to the World Health Organisation (WHO) criteria.
* Diagnosed with neuropathic pain due to distal symmetrical diabetic neuropathy of at least six months duration, as defined by a NDS score of at least 4, and in who pain is not wholly relieved with their current therapy. The NDS score must be attained from at least two different test parameters and not only the ankle jerk reflex.
* The last six daily diary 0-10 NRS pain scores before randomisation summed to at least 24.
* Stable dose of regular pain medication and non-pharmacological therapies (including TENS) for at least 14 days prior to the screening visit and willingness for these to be maintained throughout the study.
* Agreement for the responsible authorities (as applicable in individual countries), their primary care physician, and their consultant, if appropriate, to be notified of their participation in the study.

Exclusion Criteria:

* Concomitant pain thought by the investigator to be of a nature or severity to interfere with their assessment of their painful diabetic neuropathy.
* Uncontrolled diabetes with HbA1c blood levels of more than 11% at Visit1, Day B1.
* Receiving a prohibited medication and were unwilling to stop or comply for the duration of the study.
* Has used cannabinoid based medications within 60 days of study entry and were unwilling to abstain for the duration for the study.
* Has used cannabis within 30 days of study entry and were unwilling to abstain for the duration for the study.
* History of schizophrenia, other psychotic illness, severe personality disorder or other significant psychiatric disorder other than depression associated with their underlying condition.
* Known or suspected history of alcohol or substance abuse.
* History of epilepsy or recurrent seizures.
* Known or suspected hypersensitivity to cannabinoids or any of the excipients of the IMP.
* Postural drop of 20mmHg or more in systolic blood pressure at screening.
* Medical history of gastroparesis.
* Evidence of cardiomyopathy.
* Experienced myocardial infarction or clinically relevant cardiac dysfunction within the last 12 months or had a cardiac disorder that, in the opinion of the investigator would put the subject at risk of a clinically relevant arrhythmia or myocardial infarction.
* QT interval; of > 450 ms (males) or > 470 ms (females) at Visit 1.
* Secondary or tertiary AV block or sinus bradycardia (HR <50bpm) or sinus tachycardia (HR>110bpm) at Visit 1.
* Diastolic blood pressure of <50 mmHg or >105 mmHg in a sitting position at rest for five minutes prior to randomisation.
* Impaired renal function i.e., creatinine clearance is lower than 50 ml/min at Visit 1.
* Significantly impaired hepatic function, at Visit 1, in the investigator's opinion.
* Female subjects of child bearing potential and male subjects whose partner was of child bearing potential, unless they were willing to ensure that they or their partner used effective contraception during the study and for three months thereafter.
* If female, were pregnant or lactating, or were planning pregnancy during the course of the study and for three months thereafter.
* Received an IMP within the 12 weeks before Visit 1.
* Any other significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, may influence the result of the study, or the subject's ability to participate in the study.
* Following a physical exam, the subject had any abnormalities that, in the opinion of the investigator, would prevent the subject from safely participating in the study.
* Intention to donate blood during the study.
* Intention to travel internationally during the study.
* Previous randomisation into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2005-07; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Solomon Tesfaye, JCHMT FRCP, Principal Investigator — Royal Hallamshire Hospital
Locations (1):
- Royal Hallamshire Hospital, Sheffield, Yorkshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Sativex: Contains Δ9 tetrahydrocannabinol (THC), 27 mg/ml: cannabidiol (CBD), 25 mg/ml delivered in 100 microlitre actuations by a pump action oromucosal spray. Maximum permitted dose was 24 actuations (THC 65 mg: CBD 60 mg) in 24 hours
- Placebo: Contains no active drug but colourants and excipients. Maximum permitted dose was 24 actuations in 24 hours.
Period: Overall Study
Arm/Group | Sativex | Placebo
Started | 149 | 148
Completed | 105 | 125
Not Completed | 44 | 23
Not completed — Adverse Event | 30 | 12
Not completed — Lack of Efficacy | 4 | 5
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Refused medication, no side effects | 1 | 0
Not completed — Non-compliance with stable analgesia | 1 | 0
Not completed — Did not meet entry criteria at visit 1 | 1 | 0
Not completed — Subject thought medication changed | 1 | 0
Not completed — Ceased treatment due to travel | 1 | 0
Not completed — Subject preferred paracetamol | 0 | 1
Not completed — Felt good so stopped treatment | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sativex | Placebo | Total
Number analyzed (Participants) | 149 | 148 | 297
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 97 | 119 | 216
  >=65 years | 52 | 29 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (10.38) | 58.2 (10.57) | 59.5 (10.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 58 | 114
  Male | 93 | 90 | 183
Region of Enrollment [Number; unit: participants]
  United Kingdom | 91 | 86 | 177
  Czech Republic | 34 | 37 | 71
  Romania | 24 | 25 | 49

OUTCOME MEASURES:

1. Primary Outcome: The Change From Baseline in Mean Diabetic Neuropathy Pain 0-10 Numerical Rating Scale Score at the End of Treatment (Average of Last 7 Days Treatment)
Description: The diabetic neuropathy pain Numerical Rating Scale was complete at the end of every day. The patient was asked "on a scale of '0 to 10', please indicate the number that best describes your nerve pain due to diabetes in the last 24 hours" where 0 = no pain and 10 = worst possible pain. No pain relates to the time prior to the onset of pain due to diabetic neuropathy. For those whose evaluable period ended before Day 7, the mean of the available post-randomisation data was used. Those with no post-baseline diary pain 0-10 Numerical Rating Scale scores were excluded from the analysis.
Time Frame: Day 0 to Day 98
Population: The primary population for analysis was the full analysis set, which included all randomised subjects who received at least one dose of study medication and yielded on-treatment efficacy data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 146 | 148
units on a scale | -1.67 (2.13) | -1.55 (2.09)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The model used for the analysis of the end of study value was an analysis of covariance (ANCOVA) with baseline value as a covariate and treatment group and centre group as main effect. The test was performed at the 10% significance level as a possible indicator of an interactive effect. The null hypothesis was one of no difference between treatments; Test type: Superiority or Other; p = 0.634, ANCOVA; estimated treatment effect = -0.12, 95% CI 2-sided [-0.60 to 0.36] — A negative difference in treatment effect indicates an improvement in pain in favour of Sativex

2. Secondary Outcome: Change From Baseline in Mean Neuropathic Pain Scale Score at the End of Treatment
Description: The Neuropathic Pain Scale score is the 0-100 sum of 10 individual pain scores (0-10 Numerical Rating Scale, 0= no pain to 10 = most pain imaginable). A negative change from baseline indicates an improvement in pain. The baseline mean Neuropathic Pain Scale score was to be the mean of the two assessments during the baseline period, with the end of study value as the mean of the last two assessments made during the evaluable period.
Time Frame: Day 0 to Day 98
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 135 | 140
units on a scale | -13.70 (19.91) | -14.16 (17.42)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The change from baseline in mean neuropathic pain scale scale score at the end of treatment was to be compared between treatment groups using ANCOVA. The model was to include treatment and centre group as factors and baseline mean usage as a covariate; Test type: Superiority or Other; p = 0.865, ANCOVA; Estimated mean treatment difference = 0.37, 95% CI 2-sided [-3.87 to 4.61], Standard Error of Mean 2.153

3. Secondary Outcome: Change From Baseline in Mean Sleep Quality 0-10 Numerical Rating Scale Score at the End of Treatment
Description: The sleep quality Numerical Rating Scale was completed at the same time each day, i.e. bedtime in the evening. The patient was asked "on a scale of '0 to 10', please indicate the number that best describes your sleep quality in the last 24 hours" where 0 = slept extremely well and 10 = unable to sleep at all. A negative value indicates an improvement in pain score from baseline. The analyses were based on the change from baseline for the last assessment falling within the evaluable period (considered the end of treatment).
Time Frame: Day 0 - Day 98
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 132 | 142
units on a scale | -2.0 (3.02) | -1.6 (2.76)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The change from baseline in mean sleep quality numerical rating scale score at the end of treatment was compared between treatment groups using ANCOVA. The model included treatment and centre group as factors and baseline mean usage as a covariate; Test type: Superiority or Other; p = 0.139, ANCOVA; Estimated mean treatment difference = -0.45, 95% CI 2-sided [-1.04 to 0.15]

4. Secondary Outcome: Subject Global Impression of Change at the End of Treatment
Description: The subject was to assess the change in their nerve pain due to diabetic neuropathy at the end of the study compared to baseline on a 7-point scale from very much worse to very much improved. The number of participants reporting each score is presented.
Time Frame: Day 0 and Day 98
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 140 | 141
participants
  Very Much Improved | 13 | 14
  Much Improved | 40 | 36
  Slightly Improved | 48 | 35
  No Change | 30 | 45
  Slightly worse | 6 | 9
  Much worse | 2 | 2
  Very much worse | 1 | 0
Statistical Analysis 1: Comparison: Sativex vs Placebo; In the analysis of Subject Global Impression of Change, the two treatment groups were compared using ordinal logistic regression and the proportional odds model. The model incorporated centre group as a factor; Test type: Superiority or Other; p = 0.219, Regression, Logistic; Odds Ratio (OR) = 1.301, 95% CI 2-sided [0.855 to 1.981]

5. Secondary Outcome: Change From Baseline in Mean Brief Pain Inventory (Short Form)'Pain Severity Composite Score' at the End of Treatment
Description: The brief pain inventory (short form) is a 14-item questionnaire that asks patients to rate pain over the prior week and the degree to which it interferes with activities on a 0 to 10 scale, where 0=no pain and 10=pain as bad as you can imagine. Severity is measured as worst pain, least pain, average pain, and pain right now. The pain severity composite score was calculated as the arithmetic mean of the four severity items (range 0-10). The minimum value is zero and maximum is 10. A higher score represents a poor outcome.
Time Frame: Day 0 and Day 98
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 137 | 135
units on a scale | -1.2 (1.92) | -1.2 (2.06)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The change from baseline in mean brief pain inventory (short form) composite score at the end of treatment was compared between treatment groups using ANCOVA. The model included treatment and centre group as factors and baseline mean usage as a covariate; Test type: Superiority or Other; p = 0.841, ANCOVA; estimated mean treatment difference = -0.05, 95% CI 2-sided [-0.51 to 0.42]

6. Secondary Outcome: Change From Baseline in Mean Quality of Life EuroQol 5-D Weighted Health State Index Score at the End of Treatment Measured by Visual Analogue Scale
Description: The EuroQol-5D Health Status Visual Analogue Scale rated the health state on a scale of 0-100 with 0 = worst health state imaginable to 100 = best health state imaginable. An increase in score indicates an improvement in condition.
Time Frame: Day 0 and Day 98
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 138 | 135
units on a scale | 3.3 (22.26) | 7.8 (22.91)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The change from baseline in weighted health state index score at the end of treatment was compared between treatment groups using ANCOVA. The model included treatment and centre group as factors and baseline symptom score as a covariate; Test type: Superiority or Other; p = 0.523, ANCOVA; Median Difference (Final Values) = -0.01, 95% CI 2-sided [-0.06 to 0.03], Standard Error of Mean 0.021

7. Secondary Outcome: Change From Baseline in the Use of Rescue Analgesia at the End of Treatment
Description: The mean daily number of paracetamol tablets used were calculated for the periods over which the primary endpoint was calculated.
Time Frame: Day 0 - Day 98
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Tablets
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 146 | 148
Tablets | -0.53 (2.02) | -0.35 (1.94)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The model used for the analysis of the end of study value was ANCOVA with baseline value as a covariate and treatment group and centre group as main effect. The test was performed at the 10% significance level as a possible indicator of an interactive effect. The null hypothesis was one of no difference between treatments. A negative difference in adjusted means indicates an improvement in favour of Sativex; Test type: Superiority or Other; p = 0.410, ANCOVA; estimated mean treatment difference = -0.17, 95% CI 2-sided [-0.59 to 0.24]

8. Secondary Outcome: Incidence of Adverse Events as a Measure of Subject Safety
Description: The number of subjects who experienced an adverse event during the course of the study (including the follow-up period i.e 28 days after the end of treatment) is presented.
Time Frame: Day 0 - Day 133
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 149 | 148
participants
  All-causality relationship to study medication | 120 | 101
  Plausibly related to study medication | 96 | 52

9. Secondary Outcome: Change From Baseline in Mean Intoxication 0-10 Numerical Rating Scale Score at the End of Treatment
Description: Subjects rated their intoxication levels on a scale of 0-10, where 0 equals "no intoxication" and 10 equals "extreme intoxication". A negaitve value from baseline indicates and improvement. End of treatment was classed as the last on-treatment visit where data was recorded.
Time Frame: Day 0 - Day 98
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 142 | 145
units on a scale | 0.8 (2.73) | -0.3 (1.96)

10. Primary Outcome: Number of Responders at the 30% Improvement Level at the End of Treatment
Description: A positive 30% pain response is defined as a reduction of at least 30% in the mean NRS average pain score from baseline to week 14 (last 7 days). The patient was asked "on a scale of '0 to 10', please indicate the number that best describes your pain or average pain in the last 24 hours" where 0 = no pain and 10 = pain as bad as you can imagine. No pain relates to the time prior to the onset of pain. The average pain NRS was completed at the same time each day, i.e. bedtime in the evening. Estimates were produced for a one-week period, with the evaluable period finishing at the end of the appropriate seven-day period.
Time Frame: Day 0 - Day 98
Population: All subjects who were randomised and received at least one actuation of study medication were included in the analysis. Subjects with no data during the primary period (i.e. unknown response) were included in the analysis, and were classed as non-responders.
Measure: Number; unit: participants
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 149 | 148
participants | 54 | 59
Statistical Analysis 1: Comparison: Sativex vs Placebo; The numbers of responders were to be analysed using the difference in proportions and the odds ratio comparing the treatment groups with the provision of 95% CIs for the difference and odds ratio; Test type: Superiority or Other; p = 0.521, Regression, Logistic; Odds Ratio (OR) = 0.857, 95% CI 2-sided [0.537 to 1.370]

ADVERSE EVENTS:
Time Frame: All adverse events occurring from the time of consent to post study follow up i.e. 19 weeks were collected. All deaths and serious adverse events occurring within 28 days of the final dose of study medication were also collected.
Description: All adverse events occurring during the study were reported on the running logs at the back of the study case report form.
Arm/Group | Sativex | Placebo
Serious Adverse Events (participants affected / at risk) | 14/149 | 12/148
Other Adverse Events (participants affected / at risk) | 120/149 | 101/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sativex (N=149) | Placebo (N=148)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 | 0
BRADYCARDIA (Cardiac disorders) | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 1
EYE HAEMORRHAGE (Eye disorders) | 0 | 1
GASTROINTESTINAL INFLAMMATION (Gastrointestinal disorders) | 1 | 0
PERIODONTITIS (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1
GASTRITIS (Gastrointestinal disorders) | 0 | 1
HAEMATEMESIS (Gastrointestinal disorders) | 0 | 1
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 0 | 1
NAUSEA (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 0 | 1
OEDEMA PERIPHERAL (General disorders) | 0 | 1
PYREXIA (General disorders) | 0 | 1
CELLULITIS (Infections and infestations) | 1 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0
BLOOD GLUCOSE INCREASED (Investigations) | 0 | 1
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 1 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0
KETOACIDOSIS (Metabolism and nutrition disorders) | 1 | 0
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
EXOSTOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
ISCHAEMIC STROKE (Nervous system disorders) | 1 | 0
SYNCOPE (Nervous system disorders) | 1 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 0 | 1
ESSENTIAL HYPERTENSION (Vascular disorders) | 1 | 0
PERIPHERAL OCCLUSIVE DISEASE (Vascular disorders) | 1 | 0
ACCELERATED HYPERTENSION (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sativex (N=149) | Placebo (N=148)
Dizziness (Nervous system disorders) | 42 | 7
Somnolence (Nervous system disorders) | 11 | 7
Headache (Nervous system disorders) | 9 | 11
Lethargy (Nervous system disorders) | 5 | 1
Amnesia (Nervous system disorders) | 4 | 2
Dysgeusia (Nervous system disorders) | 4 | 1
Memory impairment (Nervous system disorders) | 4 | 1
Nausea (Gastrointestinal disorders) | 25 | 15
Vomiting (Gastrointestinal disorders) | 14 | 11
Dry mouth (Gastrointestinal disorders) | 12 | 4
Diarrhoea (Gastrointestinal disorders) | 10 | 14
Oral pain (Gastrointestinal disorders) | 7 | 0
Abdominal pain upper (Gastrointestinal disorders) | 5 | 2
Mouth ulceration (Gastrointestinal disorders) | 4 | 2
Oral discomfort (Gastrointestinal disorders) | 4 | 4
Fatigue (General disorders) | 10 | 4
Feeling abnormal (General disorders) | 4 | 0
Oedema peripheral (General disorders) | 4 | 2
Nasopharyngitis (Infections and infestations) | 8 | 6
Lower respiratory tract infection (Infections and infestations) | 6 | 8
Urinary tract infection (Infections and infestations) | 2 | 8
Disorientation (Psychiatric disorders) | 8 | 1
Depression (Psychiatric disorders) | 5 | 2
Insomnia (Psychiatric disorders) | 0 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 9 | 5
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 5
Palpitations (Cardiac disorders) | 4 | 1
Vertigo (Ear and labyrinth disorders) | 6 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GW will coordinate the dissemination of data from this study and may solicit input and assistance from the principal investigator. All publications, for example manuscripts, abstracts, oral/slide presentations or book chapters based on this study, must be submitted to GW for corporate review before release.